CLINICAL TRIAL: NCT06427382
Title: Prediction of Hypotension Using Perfusion Index Following Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, anesthesiology and reanimation associate professor, Ankara Yildirim Beyazıt University
Other Study IDs: perfusion index
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia, Spinal
Keywords: spinal anesthesia; perfusion index; orthopedic surgery
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group E (age > 65 years): Patients aged 65 years and older
  Interventions: Device: Perfusion index
- group N (age < 65 years): Patients aged 18 to 65 years
  Interventions: Device: Perfusion index

INTERVENTIONS:
Device: Perfusion index — Perfusion index determination using non-invasive pulse oximetry

SUMMARY:
It is aimed to investigate whether the perfusion index (PI) can predict hypotension after spinal anesthesia in elderly patients as much as in non-elderly patients.

DETAILED DESCRIPTION:
In orthopedic lower extremity surgeries, spinal anesthesia is a preferred method of anesthesia compared to general anesthesia. Spinal anesthesia may cause severe hypotension and adverse effects in the patient due to pharmacologic sympathectomy. Especially elderly patients and patients with comorbid diseases are at risk. Hypoperfusion and vasopressor drugs to be used in treatment may lead to adverse effects.

Perfusion index is calculated as the ratio non-pulsatile to pulsatile flow in peripheral capillary blood flow. Perfusion index is a non-invasive method that provides insight into the dynamics of vascular tone using pulse oximetry. It can be used to evaluate perfusion dynamics due to changes in peripheral vascular tone and to detect the possibility of developing hypotension following spinal anesthesia. There is insufficient data to assess whether PI is a marker of hypotension after spinal anesthesia in older patients compared to non-elderly patients. The planned study aims to investigate whether PI predicts hypotension after spinal anesthesia in older patients as well as non-elderly patients.

Preoperative demographic data of the patients, preoperative heart rate, noninvasive systolic, and diastolic blood pressures, mean arterial pressures, and peripheral oxygen saturations will be measured and noted. For the initial perfusion index (PI) value, PI measurements will be taken 3 times at a few minute intervals with a noninvasive probe attached to the finger, and the average will be recorded as the initial PI value. Spinal anesthesia will be applied by injecting an appropriate dose of 0.5% hyperbaric bupivacaine intrathecally, depending on the patient is structure and the type of surgery, to ensure adequate sensory and motor blockade. The patient will be immediately placed in the supine position. After the appropriate period, the level of sensory blockade will be evaluated. Heart rate, noninvasive systolic, and diastolic blood pressures, mean arterial pressure, peripheral oxygen saturation, and perfusion index will be recorded. Hypotension after spinal anesthesia will be defined as systolic blood pressure less than 90 mmHg, systolic blood pressure decrease by more than 25% from the preoperative baseline value, or average blood pressure less than 60 mmHg. Patients under the age of 65 or over the age of 65 who will undergo lower extremity surgery under spinal anesthesia will be evaluated in two groups. It will be examined whether there are differences between the groups in terms of demographic data (age, gender, comorbidity, etc.) and perfusion index.

The study's primary outcome is to investigate whether PI values have a predictive value in predicting post-spinal hypotension between the two groups and, if so, whether there is a statistically significant difference.

The secondary outcome is to evaluate whether the perfusion index can be used to predict spine-induced hypotension in orthopedic lower extremity surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II-III physical status
* patients planned for effective lower extremity surgery in the supine position
* age >18 years

Exclusion Criteria:

* Known cardiac abnormalities (left ventricular ejection fraction <50% or decompensated heart failure, heart block, arrhythmia)
* uncontrolled hypertension
* hyperthyroidism
* monoamine oxidase inhibitor use
* chronic beta-blocker or digoxin therapy
* severe arrhythmia
* peripheral arterial disease
* history of glaucoma
* hepatic cell failure
* renal failure
* local anesthetic allergy
* contraindications for spinal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients admitted to ankara city hospital for lower extremity surgery in supine position
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Perfusion index age difference | 1 hours
  Determine a threshold for baseline PI value using logistic regression analysis to predict hypotension after spinal anesthesia

SECONDARY OUTCOMES:
Perfusion index cut-off point | 1 hours
  Determining baseline perfusion index threshold to predict possible hypotension after spinal anesthesia
Systolic blood pressure | 1 hours
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the end of the procedure
Diastolic blood pressure | 1 hours
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the end of the procedure
Mean arterial pressure | 1 hours
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the end of the procedure
Hearth Rate | 1 hours
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the end of the procedure
perfusion index | 1 hours
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the end of the procedure
oxygen saturation(SpO2) | 1 hours
  recorded every 2 minutes for the first 15 minutes, then every 5 minutes until the end of the procedure
bromage score | 1 hours
  time to reach the bromage 3 score
T10 dermatome | 1 hours
  time to reach t10 dermatome level
dermatomal level | 1 hours
  the highest dermatome level achieved with spinal anesthesia
use ephedrine | 24 hours
  ephedrine use
side effects | 24 hours
  To study side effects between 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya,, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No